CLINICAL TRIAL: NCT01501929
Title: Effects of Nebivolol on Microvascular Perfusion in the Skeletal Muscles During Exercise in Hypertensive Patients
Brief Title: Effects of Nebivolol on Skeletal Muscle During Exercise in Hypertensive Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Principal Investigator, Wanpen Vongpatanasin, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: Bystolic MD52
Record Dates: First submitted 2011-11-29; First posted 2011-12-30 (Estimated); Results first posted 2018-11-06 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-05

CONDITIONS: Hypertension
Keywords: hypertension; blood pressure; blood pressure medications; metoprolol; nebivolol; vascular oxidative stress; nitric oxide; nitric oxide synthase (eNOS); endothelium; endothelial dysfunction; endothelial cell protein expression; microvascular blood flow; flow mediated dilation; handgrip exercise; endothelial cell collection; microbubbles; Definity
MeSH Terms: conditions — Hypertension | interventions — Metoprolol; Nebivolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Initial treatment with metoprolol (Active Comparator): The subject will be started on metoprolol succinate (Toprol XL) 100-300mg daily, which he/she will continue for a period of 12 weeks. Following the 12-week treatment period, the procedures listed below will be performed. After completion of the study procedures, the medication will be discontinued. If necessary, 2 weeks after drug withdrawal, subjects will be started on HCTZ if BP > 140/90 mmHg and will continue HCTZ for a 2-week period, after which the subject will be transitioned to nebivolol (Bystolic) 5-20mg daily, which he or she will continue for a period of 12 weeks. Following the 12-week treatment period, the procedures listed below will be performed. After completion of the study procedures, the medication will be discontinued.
  Interventions: Drug: Metoprolol succinate; Drug: Nebivolol; Procedure: Non-invasive measurement of Cardiac Output (CO); Procedure: Endothelial cell collection; Procedure: Microvascular perfusion assessment using Definity
- Initial treatment with nebivolol (Active Comparator): The subject will be started on nebivolol (Bystolic) 5-20mg daily, which he or she will continue for a period of 12 weeks. Following the 12-week treatment period, the procedures listed below will be performed. After completion of the study procedures, the medication will be discontinued. If necessary, 2 weeks after drug withdrawal, subject will be started on HCTZ if BP > 140/90 mmHg and will continue HCTZ for a 2-week period, after which the subject will be transitioned to metoprolol succinate (Toprol XL) 100-300mg daily, which he or she will continue for a period of 12 weeks. Following the 12-week treatment period, the procedures listed below will be performed. After completion of the study procedures, the medication will be discontinued.
  Interventions: Drug: Metoprolol succinate; Drug: Nebivolol; Procedure: Non-invasive measurement of Cardiac Output (CO); Procedure: Endothelial cell collection; Procedure: Microvascular perfusion assessment using Definity

INTERVENTIONS:
Drug: Metoprolol succinate — The subject will be started on metoprolol succinate (Toprol XL) 100-300mg daily, which he or she will continue for a period of 12 weeks. Following the 12-week treatment period, the procedures listed below will be performed. After completion of the study procedures, the medication will be discontinued.
  Other Names: Toprol XL
Drug: Nebivolol — The subject will be started on nebivolol (Bystolic) 5-20mg daily, which he or she will continue for a period of 12 weeks. Following the 12-week treatment period, the procedures listed below will be performed. After completion of the study procedures, the medication will be discontinued.
  Other Names: Bystolic
Procedure: Non-invasive measurement of Cardiac Output (CO) — Cardiac Output (CO) will be measured non-invasively at rest and during exercise by thoracic electrical bioimpedance. Stroke volume will be derived from change in impedance/time measured during electrical systole. Cardiac output will be determined as the product of stroke volume and heart rate.
  Other Names: Cardiac output by thoracic electrical bioimpedance; Bioz, Cardio Dynamics International Corporation
Procedure: Endothelial cell collection — We will collect endothelial cells from a superficial vein, usually in the arm. Following insertion of a peripheral intravenous (IV) catheter, we will collect cells from the inner lining of the vein using a thin, flexible J-tipped wire. The wire will be inserted through the IV into the vein and then removed, along with a sampling of endothelial cells. The cells collected will be processed and stained for several proteins involved in endothelial cell function, using immunofluorescent technique.
  Other Names: Endocell collection
Procedure: Microvascular perfusion assessment using Definity — Using high-resolution ultrasound, we will measure skeletal muscle blood flow during infusion of a solution containing the octafluoropropane microbubble contrast agent, Definity. The solution will be a dilution of 1 vial of Definity to 30 cc of normal saline. The ultrasound probe will be placed over the forearm to obtain images while octafluoropropane microbubbles (Definity) are infused intravenously at the rate of 0.20 to 0.27 ml/min, not to exceed a maximum dose of 2 vials per study subject per day or visit. The microvascular perfusion assessment using Definity be performed at rest as well as during slow and fast handgrip exercises.

SUMMARY:
The purpose of this study is to determine if Nebivolol improves microvascular perfusion in skeletal muscle during exercise in hypertensive patients and whether this improvement is accompanied by reduction in vascular oxidative stress or increased endothelial nitric oxide synthase (eNOS) expression in humans.

DETAILED DESCRIPTION:
In 32 untreated stage 1 hypertensive subjects, the investigators will measure blood pressure; noninvasive cardiac output by thoracic electrical bioimpedance (Bioz, Cardio Dynamics); forearm mediated vasodilation (FMD), which is a non-invasive assessment of endothelial function; collect venous endothelial cells; and measure microvascular perfusion using an Octafluoropropane microbubble contrast agent (Definity).

To obtain FMD, the brachial artery will be imaged using ultrasound. After a clear picture has been obtained, the cuff on the same arm will be inflated until it is tight for five minutes. During and following this, the subject's arm will continue to be imaged to monitor maximal increase in the brachial artery diameter.

To collect endothelial cells, a thin wire will be inserted in the vein to collect cells from the inner lining of the vein. The cells collected will be processed and stained for several proteins involved in endothelial cell function, using immunofluorescent technique.

To assess the microvascular perfusion in the skeletal muscle, a contrast agent (Definity) will be administered at baseline and after 5 minutes of rhythmic hand grip exercise at 30% of maximal voluntary contraction.

The investigators will then randomize our subjects to receive 12 weeks of Metoprolol or Nebivolol, using a cross over design. There will be a 4 week washout period between the two treatments. During the washout period, subjects will be followed after 2 weeks of drug withdrawal. Subjects found to have BP > 140/90 mmHg then, will be started on hydrochlorothiazide (HCTZ) at 25 mg once daily. Then subjects will be asked to return in 2 weeks. At that time HCTZ will be stopped if started in the earlier visit, and subject will be switched to the remaining treatment (Nebivolol or Metoprolol). Then, the investigators will assess microvascular perfusion in the skeletal muscle at rest and during handgrip exercise, endothelial function (FMD), and changes in endothelial cell protein expression after 12 weeks of Nebivolol and after 12 weeks of Metoprolol treatment in the same subjects.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with stage I primary untreated hypertension (BP between 140-159/90-99 mmHg)
* Age 18-65

Exclusion Criteria:

* Congestive heart failure
* Coronary artery disease
* Left ventricular hypertrophy by echocardiography or ECG
* History of stroke
* Average blood pressure >159/99 mmHg
* Bradycardia with a resting heart rate <55 bpm
* Chronic kidney disease with a serum creatinine > 1.4 mg/dL
* Asthma or chronic obstructive pulmonary disease
* Women who are pregnant or planning to become pregnant
* Hypersensitivity to beta blockers, hydrochlorothiazide, or Definity
* Any history of substance abuse (other than tobacco)
* Concomitant drug treatment which raises endogenous nitric oxide levels, including nitrates or phosphodiesterase V inhibitors (Viagra, Levitra)
* History of symptomatic bradycardia or heart block
* Patients with Right-to-left, bidirectional, or transient right-to-left cardiac shunts
* Hypersensitivity to perflutren, blood, blood products or albumin.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wanpen Vongpatanasin, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

REFERENCES:
- [Background] Hamada M, Kazatani Y, Shigematsu Y, Ito T, Kokubu T, Ishise S. Enhanced blood pressure response to isometric handgrip exercise in patients with essential hypertension: effects of propranolol and prazosin. J Hypertens. 1987 Jun;5(3):305-9. doi: 10.1097/00004872-198706000-00007. PMID 3302040
- [Background] Saitoh M, Miyakoda H, Kitamura H, Kinugawa T, Hisatome I, Kotake H, Mashiba H. Cardiovascular and sympathetic nervous response to dynamic exercise in patients with essential hypertension. Intern Med. 1992 May;31(5):606-10. doi: 10.2169/internalmedicine.31.606. PMID 1387013
- [Background] Glezer GA, Lediashova GA. Changes in general haemodynamics and renal function during exercise in patients with arterial hypertension. Cor Vasa. 1975;17(1):1-13. PMID 1149456
- [Background] Kazatani Y, Hamada M, Shigematsu Y, Hiwada K, Kokubu T. Beneficial Effect of a Long-Term Antihypertensive Therapy on Blood Pressure Response to Isometric Handgrip Exercise in Patients with Essential Hypertension. Am J Ther. 1995 Mar;2(3):165-169. doi: 10.1097/00045391-199503000-00003. PMID 11847547
- [Background] Marraccini P, Palombo C, Giaconi S, Michelassi C, Genovesi-Ebert A, Marabotti C, Fommei E, Ghione S, L'Abbate A. Reduced cardiovascular efficiency and increased reactivity during exercise in borderline and established hypertension. Am J Hypertens. 1989 Dec;2(12 Pt 1):913-6. doi: 10.1093/ajh/2.12.913. PMID 2610996
- [Background] Kokkinos PF, Andreas PE, Coutoulakis E, Colleran JA, Narayan P, Dotson CO, Choucair W, Farmer C, Fernhall B. Determinants of exercise blood pressure response in normotensive and hypertensive women: role of cardiorespiratory fitness. J Cardiopulm Rehabil. 2002 May-Jun;22(3):178-83. doi: 10.1097/00008483-200205000-00009. PMID 12042686
- [Background] Schutz W, Hortnagl H, Magometschnigg D. Function of the autonomic nervous system in young, untreated hypertensive patients. Int J Cardiol. 1986 Feb;10(2):133-40. doi: 10.1016/0167-5273(86)90221-4. PMID 3002992
- [Background] Goodman JM, McLaughlin PR, Plyley MJ, Holloway RM, Fell D, Logan AG, Liu PP. Impaired cardiopulmonary response to exercise in moderate hypertension. Can J Cardiol. 1992 May;8(4):363-71. PMID 1535538
- [Background] Lund-Johansen P. Twenty-year follow-up of hemodynamics in essential hypertension during rest and exercise. Hypertension. 1991 Nov;18(5 Suppl):III54-61. doi: 10.1161/01.hyp.18.5_suppl.iii54. PMID 1937687
- [Background] de Champlain J, Petrovich M, Gonzalez M, Lebeau R, Nadeau R. Abnormal cardiovascular reactivity in borderline and mild essential hypertension. Hypertension. 1991 Apr;17(4 Suppl):III22-8. doi: 10.1161/01.hyp.17.4_suppl.iii22. PMID 2013489
- [Background] Zhao W, Swanson SA, Ye J, Li X, Shelton JM, Zhang W, Thomas GD. Reactive oxygen species impair sympathetic vasoregulation in skeletal muscle in angiotensin II-dependent hypertension. Hypertension. 2006 Oct;48(4):637-43. doi: 10.1161/01.HYP.0000240347.51386.ea. Epub 2006 Aug 28. PMID 16940212
- [Background] Ladage D, Brixius K, Hoyer H, Steingen C, Wesseling A, Malan D, Bloch W, Schwinger RH. Mechanisms underlying nebivolol-induced endothelial nitric oxide synthase activation in human umbilical vein endothelial cells. Clin Exp Pharmacol Physiol. 2006 Aug;33(8):720-4. doi: 10.1111/j.1440-1681.2006.04424.x. PMID 16895546
- [Background] Reidenbach C, Schwinger RH, Steinritz D, Kehe K, Thiermann H, Klotz T, Sommer F, Bloch W, Brixius K. Nebivolol induces eNOS activation and NO-liberation in murine corpus cavernosum. Life Sci. 2007 Jun 6;80(26):2421-7. doi: 10.1016/j.lfs.2007.04.016. Epub 2007 Apr 25. PMID 17512554
- [Background] Bragadeesh T, Sari I, Pascotto M, Micari A, Kaul S, Lindner JR. Detection of peripheral vascular stenosis by assessing skeletal muscle flow reserve. J Am Coll Cardiol. 2005 Mar 1;45(5):780-5. doi: 10.1016/j.jacc.2004.11.045. PMID 15734625
- [Background] Lindner JR, Womack L, Barrett EJ, Weltman J, Price W, Harthun NL, Kaul S, Patrie JT. Limb stress-rest perfusion imaging with contrast ultrasound for the assessment of peripheral arterial disease severity. JACC Cardiovasc Imaging. 2008 May;1(3):343-50. doi: 10.1016/j.jcmg.2008.04.001. PMID 19356447
- [Background] Tzemos N, Lim PO, MacDonald TM. Nebivolol reverses endothelial dysfunction in essential hypertension: a randomized, double-blind, crossover study. Circulation. 2001 Jul 31;104(5):511-4. doi: 10.1161/hc3001.094207. PMID 11479245
- [Background] Corretti MC, Anderson TJ, Benjamin EJ, Celermajer D, Charbonneau F, Creager MA, Deanfield J, Drexler H, Gerhard-Herman M, Herrington D, Vallance P, Vita J, Vogel R; International Brachial Artery Reactivity Task Force. Guidelines for the ultrasound assessment of endothelial-dependent flow-mediated vasodilation of the brachial artery: a report of the International Brachial Artery Reactivity Task Force. J Am Coll Cardiol. 2002 Jan 16;39(2):257-65. doi: 10.1016/s0735-1097(01)01746-6. PMID 11788217
- [Background] Clerk LH, Vincent MA, Jahn LA, Liu Z, Lindner JR, Barrett EJ. Obesity blunts insulin-mediated microvascular recruitment in human forearm muscle. Diabetes. 2006 May;55(5):1436-42. doi: 10.2337/db05-1373. PMID 16644702
- [Background] Womack L, Peters D, Barrett EJ, Kaul S, Price W, Lindner JR. Abnormal skeletal muscle capillary recruitment during exercise in patients with type 2 diabetes mellitus and microvascular complications. J Am Coll Cardiol. 2009 Jun 9;53(23):2175-83. doi: 10.1016/j.jacc.2009.02.042. PMID 19497445
- [Background] Donato AJ, Gano LB, Eskurza I, Silver AE, Gates PE, Jablonski K, Seals DR. Vascular endothelial dysfunction with aging: endothelin-1 and endothelial nitric oxide synthase. Am J Physiol Heart Circ Physiol. 2009 Jul;297(1):H425-32. doi: 10.1152/ajpheart.00689.2008. Epub 2009 May 22. PMID 19465546
- [Background] Gavin KM, Seals DR, Silver AE, Moreau KL. Vascular endothelial estrogen receptor alpha is modulated by estrogen status and related to endothelial function and endothelial nitric oxide synthase in healthy women. J Clin Endocrinol Metab. 2009 Sep;94(9):3513-20. doi: 10.1210/jc.2009-0278. Epub 2009 Jun 9. PMID 19509105
- [Background] Colombo PC, Banchs JE, Celaj S, Talreja A, Lachmann J, Malla S, DuBois NB, Ashton AW, Latif F, Jorde UP, Ware JA, LeJemtel TH. Endothelial cell activation in patients with decompensated heart failure. Circulation. 2005 Jan 4;111(1):58-62. doi: 10.1161/01.CIR.0000151611.89232.3B. Epub 2004 Dec 20. PMID 15611373
- [Background] Pierce GL, Lesniewski LA, Lawson BR, Beske SD, Seals DR. Nuclear factor-kappaB activation contributes to vascular endothelial dysfunction via oxidative stress in overweight/obese middle-aged and older humans. Circulation. 2009 Mar 10;119(9):1284-92. doi: 10.1161/CIRCULATIONAHA.108.804294. Epub 2009 Feb 23. PMID 19237660
- [Derived] Velasco A, Solow E, Price A, Wang Z, Arbique D, Arbique G, Adams-Huet B, Schwedhelm E, Lindner JR, Vongpatanasin W. Differential effects of nebivolol vs. metoprolol on microvascular function in hypertensive humans. Am J Physiol Heart Circ Physiol. 2016 Jul 1;311(1):H118-24. doi: 10.1152/ajpheart.00237.2016. Epub 2016 May 13. PMID 27199121

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 32 subjects were enrolled in the study and 7 were subsequently excluded sure to various reasons, including pregnancy, normal BP of < 120/80 mmHg after the washout period of 3 week, inability to participate, and diagnosis with cancer.
Groups:
- Metoprolol First, Then Nebivolol: The subject will be started on metoprolol succinate (Toprol XL) 100-300mg daily, which he/she will continue for a period of 12 weeks. Then the subject will be switched to nebivolol (5-20 mg daily) for a period of 12 weeks.
- Nebivolol First, Then Metoprolol: The subject will be started on nebivolol (5-20 mg daily), which he/she will continue for a period of 12 weeks. Then the subject will be switched to metoprolol succinate (Toprol XL) 100-300mg daily for a period of 12 weeks.
Period: First Intervention
Arm/Group | Metoprolol First, Then Nebivolol | Nebivolol First, Then Metoprolol
Started | 8 | 17
Completed | 8 | 17
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Metoprolol First, Then Nebivolol | Nebivolol First, Then Metoprolol
Started | 8 | 17
Completed | 8 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: After the baseline measurement, all subjects were randomized to receive either nebivolol at the dose of 5 mg once daily or Metoprolol succinate 100 mg once daily, using a double-blind crossover design. If BP remained above 140/90 mmHg during the first follow-up visit, the dose of Nebivolol was increased up to 20 mg once daily and Metoprolol was increased up to 300 mg once daily.
Arm/Group | All Study Participants
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Endothelial Cell Protein Expression p47phox From Endothelial Cell Collection
Description: Endothelial cell (EC) was collected after a 20-guage angiocatheter was inserted into the contralateral forearm vein under sterile conditions. Three J-shaped vascular guidewires (St. Jude, St. Paul, MN) were advanced sequentially into the vein up to 10 cm. Endothelial cells were collected by gentle abrasion and placed into a dissociation buffer (0.5% bovine serum albumin, 2mM EDTA, and 100 ug/ml heparin in PBS). Endothelial cells were recovered from the tips of guide wires by repeated washing into collection tubes and subsequent centrifugation. EC were incubated with monoclonal antibodies against the polyclonal antibodies against NADPH oxidase p47 subunit. The intensity of staining was measured using fluorescence microscopy.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: Ratio human to HUVEC p47Phox expression
Groups:
- Metoprolol: The subject will be started on metoprolol succinate (Toprol XL) 100-300mg daily, which he/she will continue for a period of 12 weeks. The subject will be started on metoprolol succinate (Toprol XL) 100-300mg daily, which he or she will continue for a period of 12 weeks.
- Nebivolol: The subject will be started on nebivolol (Bystolic) 5-20mg daily, which he or she will continue for a period of 12 weeks.
Arm/Group | Metoprolol | Nebivolol
Number analyzed (Participants) | 25 | 25
Ratio human to HUVEC p47Phox expression | 0.47 (0.12) | 0.44 (0.07)

2. Primary Outcome: Microvascular Blood Flow
Description: Microvascular perfusion of skeletal muscle were measured during handgrip at 20 cycle per minute after 12 weeks of metoprolol, and after 12 weeks of nebivolol
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: video intensity units/ second
Arm/Group | Metoprolol | Nebivolol
Number analyzed (Participants) | 25 | 25
video intensity units/ second | 43.938 [19 to 126] | 74.584 [21 to 203]

ADVERSE EVENTS:
Groups:
- Initial Treatment With Metoprolol: The subject will be started on metoprolol succinate (Toprol XL) 100-300mg daily, which he/she will continue for a period of 12 weeks. The subject will be started on metoprolol succinate (Toprol XL) 100-300mg daily, which he or she will continue for a period of 12 weeks.
- Initial Treatment With Nebivolol: The subject will be started on nebivolol (Bystolic) 5-20mg daily, which he or she will continue for a period of 12 weeks.
Arm/Group | Initial Treatment With Metoprolol | Initial Treatment With Nebivolol
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No